CLINICAL TRIAL: NCT05390424
Title: Screening for Hepatitis B, Hepatitis C and AIDS Viruses Using Dried Blood Spot
Acronym: BUVARD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021/098/HP
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis B; Hepatitis C; AIDS
Keywords: Dried Blood Spot
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug user (Experimental): Drug users will be screened for Hepatitis C, Hepatitis B and AIDS using Dried Blood Spot for blood collection
  Interventions: Diagnostic Test: Blood collection using Dried Blood Spot

INTERVENTIONS:
Diagnostic Test: Blood collection using Dried Blood Spot — Drug users will be screened for Hepatitis C, Hepatitis B and AIDS using Dried Blood Spot for blood collection

SUMMARY:
The aim of the study is to screen for hepatitis B, hepatitis C and AIDS viruses using a Dried Blood Spot in drug users

ELIGIBILITY:
Inclusion Criteria:

* Former or active intravenous and/or nasal drug user
* Person on opiate substitution therapy

Exclusion Criteria:

* Person with known active viral infection(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Number of person with an active hepatitis C infection | Day 1
Number of person with an active hepatitis B infection | Day 1
Number of person with an active AIDS infection | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan RIACHI, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- CSAPA la Boussole, Rouen, France

IPD SHARING:
Plan to Share IPD: No